CLINICAL TRIAL: NCT00075114
Title: Promoting Self -Care to Prevent Urinary Incontinence
Brief Title: Prevent Inability To Control Urination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Carolyn Sampselle, Carolyne K. Davis Professor of Nursing, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R01NR007618-01 (NIH); R01NR007618 (NIH)
Record Dates: First submitted 2004-01-02; First posted 2004-01-05 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Urinary Incontinence
Keywords: Self Care; Behavior Modification
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Bladder Health Class (Other): A two-hour bladder health class presented by two experts in urinary incontinence and followed by an individual follow-up teaching session with an incontinence nurse specialist.
  Interventions: Behavioral: Bladder Health Class
- 2 Control Group (No Intervention): Participants randomized to this arm did not receive any interventions.

INTERVENTIONS:
Behavioral: Bladder Health Class — A two-hour bladder health class presented by two experts in urinary incontinence and followed by an individual follow-up teaching session with an incontinence nurse specialist.
  Arms: 1 Bladder Health Class

SUMMARY:
The purpose of this study is to determine the capacity of self-efficacy to predict maintaining a behavior change at four years post urinary control intervention.

DETAILED DESCRIPTION:
This is a study that will monitor and compare attitudes and strategies that women use to maintain behavior changes that prevent urination problems. Women will complete questionnaires, do muscle strength exercises, and bladder training at 3 months, one year, and 4 years post intervention.

ELIGIBILITY:
Inclusion and exclusion criteria

1. Female 55 through 80 years old
2. Post-menopausal-no menstrual cycle for the past 12 months except for women who are on hormone replacement therapy.
3. Continent of urine (using the MESA definition of continence) defined as:

   1. No previous incontinence episode except during pregnancy and/or postpartum period.
   2. Urine loss less than 6 days during the last 365 days
   3. No previous or present incontinence treatment with pharmacological agents, behavioral programs or surgical therapy.
4. No history of bladder cancer, stroke, multiple sclerosis, parkinsonism, epilepsy, spinal cord tumor or trauma.
5. No reported difficulty with activities of daily living, i.e. walking about the house, dressing, getting in/out of bed, getting to/using the toilet, bathing/showering, or eating.

Additional criteria are applied at a physical examination:

1. Mini Mental Status of at least 24
2. Negative for objective urine loss during coughing.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2000-09; Primary Completion 2002-02 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Mean number of incontinence episodes | Baseline, 6-, 12-, 18-, 24-, 32-, 42-, 48-months post baseline

SECONDARY OUTCOMES:
Pelvic floor muscle strength | Baseline, 6-, 12-, 18-, 24-, 32-, 42-, 48-months post baseline
Length of voiding interval | Baseline, 6-, 12-, 18-, 24-, 32-, 42-, 48-months post baseline
Self-efficacy | Baseline, 6-, 12-, 18-, 24-, 32-, 42-, 48-months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn M Sampselle, PhD, APH, Principal Investigator — University of Michigan, School of Nursing, MICHIN Center
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598